CLINICAL TRIAL: NCT03288389
Title: Membrane Lipid Replacement in Fibromyalgia
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: until further notice due to COVID-19 pandemic.
Sponsor: Institute for Molecular Medicine (Other)
Responsible Party: Principal Investigator, Garth Nicolson, PhD, MD (H), President & Chief Scientific Officer, Institute for Molecular Medicine
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017/02/1
Record Dates: First submitted 2017-09-13; First posted 2017-09-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Fibromyalgia
Keywords: Membrane Lipid Replacement; NTFactor Lipids; Fibromyalgia; Pain; Fatigue; Gastrointestinal symptoms
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to determine the clinical effectiveness of an all-natural, patented, Food and Drug Administration (FDA)-approved oral lipid nutritional supplement (NTFactor Lipids) on reducing pain, fatigue and other symptoms and improving quality of life in Fibromyalgia and other related conditions. The investigators will evaluate the efficacy of a dietary product called NTFactor Lipids made by Nutritional Therapeutics, Inc. of New York on pain, fatigue and gastrointestinal symptoms as well as quality of life indicators in adult male and female subjects. The addition of NTFactor Lipids to the diet is expected to improve cellular energy function, decrease fatigue and pain and lower the severity of other symptoms and improve quality of life indicators in Fibromyalgia patients. This study will be a randomized, placebo-controlled, cross-over study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomized by a nurse consultant into placebo and supplement arms and will be masked from lead investigator, physician participants and research nurse coordinator. Placebo and Product will be in identical white numbered bottles and look, feel, taste and smell the same. Data will be collected independently online by a specialty company and after the trial is completed, it will be transferred to an independent statistical unit at the University of California, Irvine for analysis and at that time the code will be broken for analysis purposes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will take 4 placebo wafers per day for 42 days. Subjects will be asked to take the Fibromyalgia Combined Symptom Survey (see attachments, based on validated survey instruments) on-line on Day 0 (before starting supplement/placebo) and on Days 1, 2, 3, 7, 14, 21, 30 and 42.
  Interventions: Dietary Supplement: Placebo
- NTFactor Lipids® (Active Comparator): Participants will take 4 NTFactor Lipid® wafers (4 g) per day for 42 days. Subjects will be asked to take the Fibromyalgia Combined Symptom Survey (see attachments, based on validated survey instruments) on-line on Day 0 (before starting supplement/placebo) and on Days 1, 2, 3, 7, 14, 21, 30 and 42.
  Interventions: Dietary Supplement: NTFactor Lipids®

INTERVENTIONS:
Dietary Supplement: NTFactor Lipids® — Membrane Lipid Replacement with NTFactor Lipids wafers
  Other Names: Patented Energy wafers
  Arms: NTFactor Lipids®
Dietary Supplement: Placebo — Placebo wafers
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the clinical effectiveness of an all-natural, patented wafer with active ingredients that are FDA approved as Generally Recognized as Safe (GRAS) Reference: US Federal Drug Administration (1970) Scientific Literature Reviews GRAS Report, PB-241 970. Active Ingredients: Lecithins. .In this study the investigators will evaluate the efficacy of this dietary product called NTFactor Lipids® made by Nutritional Therapeutics, Inc. of New York on pain, fatigue and gastrointestinal symptoms as well as quality of life indicators in adult male and female participants with fibromyalgia. The addition of NTFactor Lipids to the diet is expected to improve cellular energy function, decrease fatigue and pain and lower the severity of other symptoms and improve quality of life indicators in Fibromyalgia. This study will be a randomized, placebo-controlled, cross-over study.

DETAILED DESCRIPTION:
Adult male and female volunteers (n=60, aged 18-64) with a diagnosis of Fibromyalgia will be recruited by referral, newspapers, flyers, radio and internet ads, and asked to complete an Informed Consent document and take an on-line, validated, Combined Fibromyalgia Symptom Questionnaire or Survey Form. Potentially eligible participants (Since there are approx. twice as many female as male patients with this diagnosis, the investigators anticipate that more female than male participants will be recruited) will have the Fibromyalgia diagnosis confirmed using the American College of Rheumatology criteria. If participants have not done so, participants will be asked to provide 10 cc of blood for a Chem 20 analysis. Participants that meet the inclusion criteria will be randomized into placebo (42 days) or supplement arms (4 g NTFactor Lipids® per day for 42 days) by a Research Nurse/Associate, and blinded to the Principal Investigators and Participants for this cross-over trial. After the first arm is completed, participants will return for a clinic visit and enter the second arm for 42 days after a 2-week wash-out period. Once the data has been collected online (at Day 0 before starting supplement/placebo and on Days 1, 2, 3, 7, 14, 21, 30 and 42 for each arm), data will be placed into spread sheets, unblinded and analyzed by an independent statistical unit at the University of California, Irvine, School of Medicine. Principal objectives will be to assess various categories of pain, fatigue, GI symptoms and QOL and compare these outcomes in this study among supplement and placebo arms for each participant over time and combined for all participants. Statistical significance of any differences will be determined by t-test and other methods. Regression analysis of the data will be used to assess fidelity of the data and reliability of outcomes, and R2 values will be calculated for combined data.

ELIGIBILITY:
Inclusion Criteria:

1. You are an adult male or female (aged 18-70).
2. You have Fibromyalgia or a related clinical condition.
3. You are mobile during the day.
4. You are willing to sign an informed consent document.
5. You are willing to have 10 cc (two teaspoons) of blood drawn for analysis.
6. You are willing to take part in a clinical study that will last 14 weeks.
7. You have internet access and an email address.

Exclusion Criteria:

1. You are not an adult.
2. You do not have Fibromyalgia or a related clinical condition.
3. You are not mobile, spending more than 10 hours per day in bed.
4. You are not willing and able to sign an informed consent document.
5. You are not able to be present at a test location or have a blood draw of 10 cc (2 teaspoons) for blood analysis.
6. You have unusually high or low values on your blood chemistry screen.
7. You are pregnant
8. You have been declared mentally incompetent by a qualified health care professional.
9. You have a positive diagnosis of cancer, HIV, hepatitis and other major illnesses, such as severe hypertension, neurodegenerative or autoimmune disease.
10. You on immune suppressing drugs or medications.
11. You are legally barred from signing and informed consent document.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue as assessed by validated survey form | through study completion at 14 weeks
  Fatigue elements and overall fatigue will be self reported ten times in each six week phase
Pain as assessed by validated survey form | through study completion at 14 weeks
  Pain elements will be self reported ten times in each six week phase
Gastrointestinal symptoms as assessed by validated survey form | through study completion at 14 weeks
  Gastrointestinal symptoms will be self reported ten times in each six week phase

SECONDARY OUTCOMES:
Quality of Life as assessed by validated survey form | through study completion at 14 weeks
  QOL elements will be self reported ten times in each six week phase

CONTACTS AND LOCATIONS:
Overall Officials: Nancy C Russell, DrPH, Study Director — Independent Research Coordinator
Locations (3):
- United States (3):
  - Priority Health & Wellness, Pearland, Texas
  - Office of Dr. Paul Breeding, San Antonio, Texas
  - Blue Hole Wellness, Wimberley, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nicolson GL, Ash ME. Membrane Lipid Replacement for chronic illnesses, aging and cancer using oral glycerolphospholipid formulations with fructooligosaccharides to restore phospholipid function in cellular membranes, organelles, cells and tissues. Biochim Biophys Acta Biomembr. 2017 Sep;1859(9 Pt B):1704-1724. doi: 10.1016/j.bbamem.2017.04.013. Epub 2017 Apr 18. PMID 28432031
- [Result] Nicolson GL, Rosenblatt S, de Mattos GF, Settineri R, Breeding PC, Ellithorpe RR, Ash ME. Clinical Uses of Membrane Lipid Replacement Supplements in Restoring Membrane Function and Reducing Fatigue in Chronic Diseases and Cancer. Discoveries (Craiova). 2016 Feb 18;4(1):e54. doi: 10.15190/d.2016.1. PMID 32309576
- [Result] Nicolson GL. Mitochondrial Dysfunction and Chronic Disease: Treatment With Natural Supplements. Integr Med (Encinitas). 2014 Aug;13(4):35-43. PMID 26770107
- [Result] Nicolson GL. Membrane Lipid Replacement: clinical studies using a natural medicine approach to restoring membrane function and improving health. International Journal of Clinical Medicine 7: 133-143, 2016;